CLINICAL TRIAL: NCT07207304
Title: Evaluation Of The Influence Of Anesthetic Interventions On The Evolution Of Hepatic Neoplastic Processes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Șargarovschi Sergiu, Assistant professor, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEP45/22.11.2021
Record Dates: First submitted 2025-07-07; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: Hepato-cellular Carcinoma; Neutrophil Extracellular Trap Formation; Anesthesia; Lidocaine Infusion
Keywords: Anesthesia; Lidocaine infusion; Neutrophil Extracellular traps; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Anesthesia; Transcobalamins; Fentanyl; Analgesics, Non-Narcotic; Morphine; Consciousness Monitors; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Formation of four study groups, each around of 50 patients diagnosed with hepatocellular carcinoma or hepatic metastases, according to the type of anesthesia administered during surgery:
  Group 1 - TIVA (propofol) + lidocaine Group 2 - TIVA (propofol) + placebo Group 3 - Sevoflurane + lidocaine Group 4 - Sevoflurane + placebo
Masking Description: The laboratory physician who processed the samples was blinded to the group assignment of each sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hepatocellular carcinoma (HCC) resection performed under total intravenous anesthesia (TIVA) (Active Comparator): Patients will receive total intravenous anesthesia (TIVA) with 1% propofol, administered using the Schneider pharmacokinetic model. The initial target effect-site concentration will be 4 µg/mL, titrated intraoperatively to maintain a BIS value between 40 and 59.
  Interventions: Procedure: Anesthesia; Procedure: Anesthesia induction with TCI; Drug: Intraoperative analgesia; Drug: Non-opioid analgesics; Drug: Morphine (+); Device: Bispectral Index (BIS); Procedure: Intraoperative mechanical ventilation; Procedure: Blood sampling
- HCC resection performed under sevoflurane anesthesia (Active Comparator): Patients will receive volatile anesthesia with sevoflurane, maintained at an end-tidal concentration (EtSevo) corresponding to 1.0-1.5 MAC. The concentration will be adjusted in increments or decrements of 0.25-0.5 MAC to maintain a BIS value between 40 and 59.
  Interventions: Procedure: Anesthesia; Procedure: sevoflurane anesthesia; Drug: Intraoperative analgesia; Drug: Non-opioid analgesics; Drug: Morphine (+); Device: Bispectral Index (BIS); Procedure: Intraoperative mechanical ventilation; Procedure: Blood sampling
- HCC resection performed under TIVA + Lidocaine infusion (Active Comparator): Patients in this group will receive TIVA with 1% propofol administered via TCI using the Schneider pharmacokinetic model. A 1.5 mg/kg intravenous bolus of 1% lidocaine will be administered at induction. Following intubation, a continuous infusion of 1% lidocaine at 2 mg/kg/hour will be maintained until emergence from anesthesia, not exceeding a maximum dose of 200 mg/hour.
  Interventions: Procedure: Anesthesia; Procedure: Anesthesia induction with TCI; Drug: Lidocaine Infusion; Drug: Intraoperative analgesia; Drug: Non-opioid analgesics; Drug: Morphine (+); Device: Bispectral Index (BIS); Procedure: Intraoperative mechanical ventilation; Procedure: Blood sampling
- HCC resection performed under sevoflurane anesthesia + Lidocaine infusion (Active Comparator): Patients in this group will receive sevoflurane-based general anesthesia. Anesthesia will be maintained with sevoflurane at an end-tidal concentration of 1.0-1.5 MAC, titrated in increments or decrements of 0.25-0.5 MAC based on BIS monitoring (target range 40-59). A 1.5 mg/kg intravenous bolus of 1% lidocaine will be administered at induction, followed by a continuous intravenous infusion of 1% lidocaine at 2 mg/kg/hour, not exceeding 200 mg/hour, until emergence from anesthesia.
  Interventions: Procedure: Anesthesia; Procedure: sevoflurane anesthesia; Drug: Lidocaine Infusion; Drug: Intraoperative analgesia; Drug: Non-opioid analgesics; Drug: Morphine (+); Device: Bispectral Index (BIS); Procedure: Intraoperative mechanical ventilation; Procedure: Blood sampling

INTERVENTIONS:
Procedure: Anesthesia — Patients diagnosed with hepatocellular carcinoma will be randomly assigned to one of four groups. They will receive standard anesthesia with maintenance based on either sevoflurane or propofol. Two of the groups will additionally receive intravenous lidocaine, administered from induction until the end of surgery. Blood samples will be collected preoperatively and six hours postoperatively to measure citrullinated histone H3 (H3Cit), a reliable biomarker of NETosis. Additional inflammatory markers will also be analyzed. All patients will be followed for a period of one year
Procedure: Anesthesia induction with TCI — During induction, patients will receive fentanyl (2-3 µg/kg), propofol (1-1.5 mg/kg) as a bolus or via TCI, and rocuronium (0.5-0.6 mg/kg) to facilitate anesthesia induction and ensure adequate neuromuscular relaxation for endotracheal intubation. Anesthesia will be maintained using TIVA with 1% propofol administered via TCI, guided by the Schneider pharmacokinetic model. The initial target effect-site concentration will be 4 µg/mL and will be titrated intraoperatively to maintain a BIS value between 40 and 59.
  Arms: HCC resection performed under TIVA + Lidocaine infusion; Hepatocellular carcinoma (HCC) resection performed under total intravenous anesthesia (TIVA)
Procedure: sevoflurane anesthesia — During induction, patients will receive fentanyl (2-3 µg/kg), propofol (1-1.5 mg/kg), and rocuronium (0.5-0.6 mg/kg) to facilitate anesthesia induction and ensure adequate neuromuscular relaxation for endotracheal intubation.
  For patients in the inhalation anesthesia group, maintenance will be performed using sevoflurane. The end-tidal concentration of sevoflurane (EtSevo) will be maintained between 1.0 and 1.5 MAC, with adjustments in increments or decrements of 0.25-0.5 MAC, depending on the BIS value, which will be maintained between 40 and 59.
  Arms: HCC resection performed under sevoflurane anesthesia; HCC resection performed under sevoflurane anesthesia + Lidocaine infusion
Drug: Lidocaine Infusion — During induction, a 1.5 mg/kg intravenous bolus of 1% lidocaine will also be administered. In the maintenance phase of anesthesia, a continuous infusion of 1% lidocaine at 2 mg/kg/hour-up to a maximum of 200 mg/hour-will be administered, starting after endotracheal intubation and continued until emergence from anesthesia.
  Arms: HCC resection performed under TIVA + Lidocaine infusion; HCC resection performed under sevoflurane anesthesia + Lidocaine infusion
Drug: Intraoperative analgesia — Intraoperative analgesia will be ensured by administering fentanyl 0.5-1 µg/kg as needed, based on clinical signs of inadequate analgesia (e.g., an increase in blood pressure or heart rate exceeding 20% of baseline, mydriasis, lacrimation, or diaphoresis)
  Other Names: Fentanyl
Drug: Non-opioid analgesics — Thirty minutes before the end of surgery, nefopam 40 mg, paracetamol 1 g, and ketoprofen 100 mg will be administered intravenously, depending on the patient's comorbidities, surgical particularities, extent of resection, and residual liver volume.
Drug: Morphine (+) — Postoperative analgesia will be provided with morphine at a dose of 0.1-0.2 mg/kg, administered 30 minutes before emergence from anesthesia. The administration will be performed intravenously, with the dose adjusted based on patient weight and clinical condition. Additional bolus doses may be given in the post-anesthesia care unit (PACU), guided by the patient's reported pain intensity using the Visual Analog Scale (VAS). In the PACU, morphine will be titrated starting with 2-5 mg IV given slowly over 4-5 minutes, with repeated doses every 5-10 minutes if needed, while closely monitoring respiratory rate, level of consciousness, and hemodynamic stability. For ongoing pain management, intermittent IV bolus dosing (typically 0.05-0.1 mg/kg every 4 hours as required) may be used, taking into account factors such as patient comorbidities, type of surgery, and residual hepatic function.
Device: Bispectral Index (BIS) — Bispectral index (BIS) monitoring will be used to guide the depth of anesthesia. The target BIS value will be maintained between 40 and 59 throughout the procedure to ensure adequate hypnosis while avoiding excessive anesthetic depth. BIS values will be continuously recorded and adjustments to anesthetic agents will be made accordingly.
Procedure: Intraoperative mechanical ventilation — Intraoperative mechanical ventilation will be performed using a lung-protective strategy. Patients will be ventilated with a volume-controlled mode, using a tidal volume of 6-8 mL/kg of predicted body weight, a respiratory rate adjusted to maintain end-tidal CO₂ (EtCO₂) between 35-45 mmHg, and a positive end-expiratory pressure (PEEP) of minimum 6 cmH₂O. Fraction of inspired oxygen (FiO₂) will be set to maintain peripheral oxygen saturation (SpO₂) above 94%. Recruitment maneuvers may be applied periodically or as clinically indicated.
Procedure: Blood sampling — A total of 10 mL of peripheral venous blood will be collected from each patient at two time points: preoperatively (baseline) and 6 hours after surgery. These samples will be used to quantify the concentration of neutrophil extracellular trap (NET)-associated biomarkers, including myeloperoxidase-DNA complexes (MPO-DNA) and cell-free DNA (cfDNA), which are closely associated with NET formation. Following collection, samples will be centrifuged at 1000 rpm, and the resulting plasma will be aliquoted and stored at -80 °C for later analysis. In parallel, additional inflammatory and metabolic markers will be measured, including C-reactive protein (CRP), total leukocyte count, blood glucose, procalcitonin, and interleukin levels (IL-6, IL-8, IL-10, and IL-17) in selected patients. All participants will be monitored for a period of one year to assess the incidence of postoperative complications and cancer recurrence, including metastasis.

SUMMARY:
Evaluation Of The Influence Of Anesthetic Interventions On The Evolution Of Hepatic Neoplastic Processes

The goal of this clinical trial is to evaluate of the involvement of Neutrophil extracellular traps in the evolution of hepatocellular cancer. The main questions it aims to answer are:

* How does the type of anesthesia used in hepatobiliary oncological surgery influence postoperative evolution and the immune response?
* How does the type of anesthesia, TIVA versus inhalational influence the generation of neutrophil extracellular traps (NETs)? Researchers will compare the evolution of the patients assigned to 4 study groups depending on the anesthetic intervention performed.

Participants will:

* will be evaluated pre and postanesthesia, blood samples will be collected for analysis of the inflammatory response
* will be followed up one year for establishing the outcome

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) remains a leading cause of cancer-related mortality worldwide, with rising incidence in the context of chronic liver disease, viral hepatitis, non-alcoholic fatty liver disease, and cirrhosis. Surgical resection, whether curative or cytoreductive, is a cornerstone of management in selected patients with HCC or secondary hepatic malignancies. However, accumulating evidence highlights that perioperative factors, especially those related to anesthetic management may influence not only immediate postoperative recovery but also long-term oncologic outcomes. Debates persist regarding the optimal anesthesia for oncologic patients. While some studies favored total intravenous anesthesia (TIVA), recent retrospective studies show no significant difference between inhalational and intravenous techniques. However, adjunct therapies, such as perioperative lidocaine, may influence recurrence and outcomes.

Recent investigations into cancer biology have emphasized the role of systemic inflammation, immune dysregulation, and neutrophil behavior in promoting tumor progression, immune escape, and metastatic dissemination. A novel contributor to this inflammatory pro-tumorigenic environment is NETosis, the formation of neutrophil extracellular traps (NETs). NETs are composed of chromatin fibers (e.g., MPO, elastase, citrullinated histones), which, beyond their physiological role in infection containment, are increasingly implicated in cancer-related processes such as angiogenesis, tumor invasion, thrombosis, and immune suppression.

Research goal The aim of the study is to evaluate the involvement of NETosis in the progression of hepatocellular carcinoma.

Main objective:

To assess the influence of the type of anesthesia used in hepatobiliary oncologic surgery on postoperative evolution and immune response.

Secondary objective:

* To evaluate the impact of anesthesia type-TIVA versus inhalational-on NET formation.
* To assess the role of NETs in the progression of neoplastic disease and correlate their levels with clinical outcomes.
* To evaluate the effect of perioperative lidocaine administration on the generation of NETs.

Study type: prospective, interventional, longitudinal, randomized Methodology - presentation of work protocols

1. Logistical organization stage - ethics committee agreement; includes identification of laboratories and methods of collecting biological products (blood) for plasma concentration measurements, study-specific forms (informed consent form, data culture form)
2. Patient Enrollment Phase and Completion of Study Groups:

   2.1 Formation of four study groups, each around of 50 patients diagnosed with hepatocellular carcinoma or hepatic metastases, according to the type of anesthesia administered during surgery: Group 1 - TIVA (propofol) + lidocaine Group 2 - TIVA (propofol) + placebo Group 3 - Sevoflurane + lidocaine Group 4 - Sevoflurane + placebo

   2.2 Inclusion Criteria: Patients eligible for the study are those aged between 18 and 80 years, diagnosed with hepatocellular carcinoma or hepatic metastases, and scheduled for elective surgery (hepatectomy or metastasectomy).

   2.3 Exclusion Criteria: The following patients will be excluded from the study: those undergoing emergency surgery; patients on chronic immunosuppressive therapy; individuals with contraindications to any of the study medications; patients with psychiatric disorders (depression, bipolar disorder, schizophrenia); individuals with autoimmune diseases or corticosteroid-dependent bronchial asthma; patients with congenital or acquired coagulation disorders; chronic users of anticoagulants and/or antiplatelet agents; HIV-positive patients; pregnant women; and those receiving antiarrhythmic therapy (verapamil, propafenone, amiodarone) that may interfere with lidocaine's antiarrhythmic action.
3. Biological Sample Analysis for NETosis Quantification To quantify NETosis (which cannot be measured directly), surrogate biomarkers will be used that correlate reliably with NET formation. Promising markers include MPO-DNA complexes, cell-free DNA (cfDNA), and citrullinated histone H3 (H3Cit), all of which reflect the extent of NET generation.
4. Patient Follow-Up Patients will be followed for one year to assess overall survival and progression-free survival. Follow-up methods will include direct contact, telephone, and email. Data will be collected regarding general health status, disease progression, timing and presence of tumor recurrence, and any hospitalizations occurring after the surgical intervention along with the reasons for medical visits. Results of follow-up investigations (CT, ultrasound, and laboratory tests) requested by the attending surgeon or oncologist will be collected.
5. Data Processing and Study Completion

5.1 Analysis of H3Cit, MPO-DNA, and cfDNA concentrations in correlation with the type of anesthesia and surgical technique used.

5.2 Evaluation of associations between conventional inflammatory markers and progression of hepatocellular carcinoma or hepatic metastases.

5.3 Determination of the type of correlation between inflammatory markers and NETosis.

5.4 Comparison of plasma concentrations of local anesthetics with values reported in the literature (where antineoplastic effects were observed).

5.5 Statistical analysis and establishment of correlations between the local anesthetic used and cancer recurrence.

Brief Description of Study Procedures This is a prospective, randomized, interventional, single-center clinical trial including patients with hepatocellular carcinoma or hepatic metastases undergoing elective surgery. Tumor staging will be performed according to AJCC (American Joint Committee on Cancer) and BCLC (Barcelona Clinic Liver Cancer) criteria. Patients with ASA physical status I, II, or III will be included. Ethics approvals will be obtained from the UMF Cluj and IRGH Ethics Committees. All participants will sign written informed consent.

Inclusion criteria:

Patients aged 18-80 years with hepatocellular carcinoma or hepatic metastases undergoing elective liver resection (hepatectomy or metastasectomy).

Exclusion criteria:

Patients undergoing emergency surgery; chronic immunosuppressive therapy users; individuals with contraindications to any of the study medications; patients with psychiatric disorders (depression, bipolar disorder, schizophrenia); individuals with autoimmune diseases or corticosteroid-dependent bronchial asthma; patients with congenital or acquired coagulation disorders; chronic users of anticoagulants and/or antiplatelet agents; HIV-positive individuals; pregnant women; and patients on antiarrhythmic drugs (verapamil, propafenone, amiodarone) that could interfere with lidocaine's antiarrhythmic action.

Anesthetic protocol:

Low molecular weight heparin will be administered 12 hours prior to surgery, along with preoperative fasting as per recommendations. Premedication will include midazolam 1 mg IV. Induction will consist of fentanyl 2-3 mcg/kg, propofol 1-1.5 mg/kg, and rocuronium 0.5-0.6 mg/kg for muscle relaxation. Lidocaine 1% at 1.5 mg/kg IV bolus will also be administered at induction.

Maintenance of anesthesia:

Inhalational group: Sevoflurane administered at an EtSevo of 1-1.5 MAC, adjusted in steps of 0.25-0.5 MAC depending on BIS levels (target range 40-59).

TIVA group: Propofol administered using the Schneider pharmacokinetic model, starting with an effect-site concentration of 4 µg/ml, adjusted according to BIS (target 40-59).

All patients will receive mechanical ventilation with volume- or pressure-controlled modes, FiO₂ of 40-60% to maintain SpO₂ ≥94%, in a semi-closed circuit, with a fresh gas flow of 2-2.5 L/min, tidal volume of 6-7 mL/kg ideal body weight, and PEEP adjusted based on patient and surgical specifics.

Intraoperative analgesia:

Administer fentanyl 0.5-1 µg/kg as needed (e.g., if blood pressure or heart rate increases >20% from baseline, or signs of sympathetic activation such as mydriasis, lacrimation, sweating).

Thirty minutes before the end of surgery, nefopam 40 mg and ketoprofen 100 mg IV will be administered, depending on comorbidities.

Lidocaine infusion:

A continuous infusion of 1% lidocaine at 2 mg/kg/hour will be administered intraoperatively, up to a maximum of 200 mg/hour, from intubation until awakening.

Postoperative analgesia:

Morphine at 0.1-0.2 mg/kg IV will be administered 30 minutes prior to awakening from anesthesia.

Intraoperative monitoring:

Standard ASA monitoring (blood pressure, heart rate, temperature, peripheral oxygen saturation, end-tidal CO₂), BIS (target 40-55), and total fentanyl and lidocaine consumption will be recorded.

Blood sampling:

10 mL of peripheral venous blood will be collected preoperatively and 6 hours postoperatively to determine the levels of MPO-DNA and cfDNA, both strongly correlated with NETosis. Samples will be centrifuged at 1000 rpm, and plasma stored at -80°C. Additional inflammatory markers will be measured, including C-reactive protein (CRP), total leukocyte count, blood glucose, procalcitonin, and interleukins IL-6, IL-8, IL-10, and IL-17 for selected cases.

Patients will be followed for one year to monitor the incidence of metastases and postoperative complications.

Ethical Considerations All patients will be enrolled based on written informed consent and will be monitored according to the Research Ethics Guidelines of the "Iuliu Hațieganu" University of Medicine and Pharmacy, as well as the recommendations and requirements of the Research Ethics Committee, in compliance with international regulations and human rights protections.

The study will be approved by the Ethics Committees of UMF Cluj and IRGH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with: hepatocellular carcinoma, or hepatic metastases
* Scheduled for elective liver surgery:

Exclusion Criteria:

* Undergoing emergency surgery
* Receiving chronic immunosuppressive therapy
* Having contraindications to any of the study medications
* Diagnosed with psychiatric disorders, such as: depression, bipolar disorder, schizophrenia, having autoimmune diseases
* Suffering from corticosteroid-dependent bronchial asthma
* Diagnosed with congenital or acquired coagulation disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Survival outcomes after hepatocellular carcinoma resection. | one year postoperatively
  Patients will be followed for a period of one year to assess overall survival and progression-free survival. Follow-up will be conducted via direct contact, telephone, or e-mail. Information will be collected regarding the patient's general health status, disease progression, the presence and timing of tumor recurrence, as well as any hospitalizations occurring postoperatively, including the reason for medical consultation. Additionally, results from relevant investigations-such as computed tomography (CT), ultrasound, and blood tests-recommended by the treating surgeon or oncologist will be requested and reviewed.
NETosis quantification | Preoperatively and after 6 hours postoperatively
  For each patient, 10 mL of blood will be collected from a peripheral vein both preoperatively and 6 hours postoperatively to determine the concentrations of MPO-DNA (myeloperoxidase-DNA complexes), H3Cit (citrullinated histone H3), and cfDNA (cell-free DNA). These biomarkers are closely associated with the formation of neutrophil extracellular traps (NETs). We aim to analyze the potential relationship between the dynamics of NETosis formation, the duration of anesthesia, and postoperative patient outcomes.

SECONDARY OUTCOMES:
Quantification of the inflammatory response | Preoperatively and at 6, 12, and 24 hours postoperatively
  Samples will be collected for the analysis of inflammatory markers, C-reactive protein (CRP), total leukocyte count, blood glucose levels, and procalcitonin will be evaluated. In selected cases, interleukin levels (IL-6, IL-8, IL-10, and IL-17) will also be measured. We will analyze the relationship between the dynamics of classical inflammatory markers and NETosis across the four patient groups.
Opioid use | In the first 24 hours postoperatively
  We will evaluate the intraoperative and early postoperative opioid requirements by recording the total amount of opioids administered during surgery and in the first 24 hours postoperatively. In the initial analysis, we will compare the opioid consumption between patients who received continuous intravenous lidocaine infusion and those who did not, irrespective of the anesthetic technique used. Subsequently, we will assess potential differences in opioid requirements across all four study groups.
Length of hospital stay | From the immediate postoperative period until discharge
  We will analyze whether differences in the length of hospital stay are associated with perioperative factors such as the type of anesthesia administered, the total intraoperative and early postoperative opioid consumption, and specific surgical characteristics, including the extent of liver resection and intraoperative complications. Additionally, we will assess the impact of early postoperative events-such as the incidence of postoperative delirium, postoperative nausea and vomiting (PONV), impaired mobilization due to inadequate pain control, and opioid-related adverse effects-on prolonged hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Institute of Gastroenterology and Hepatology Octavian Fodor, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tohme S, Yazdani HO, Al-Khafaji AB, Chidi AP, Loughran P, Mowen K, Wang Y, Simmons RL, Huang H, Tsung A. Neutrophil Extracellular Traps Promote the Development and Progression of Liver Metastases after Surgical Stress. Cancer Res. 2016 Mar 15;76(6):1367-80. doi: 10.1158/0008-5472.CAN-15-1591. Epub 2016 Jan 12. PMID 26759232
- [Background] Zhao H, Wu L, Yan G, Chen Y, Zhou M, Wu Y, Li Y. Inflammation and tumor progression: signaling pathways and targeted intervention. Signal Transduct Target Ther. 2021 Jul 12;6(1):263. doi: 10.1038/s41392-021-00658-5. PMID 34248142
- [Background] Zhang W, Liu J, Li X, Bai Z, Sun Y, Chen X. Lidocaine effects on neutrophil extracellular trapping and angiogenesis biomarkers in postoperative breast cancer patients with different anesthesia methods: a prospective, randomized trial. BMC Anesthesiol. 2024 Apr 27;24(1):162. doi: 10.1186/s12871-024-02540-7. PMID 38678209
- [Background] Cata JP, Sood AK, Eltzschig HK. Anesthetic Drugs and Cancer Progression. Anesthesiology. 2020 Oct 1;133(4):698-699. doi: 10.1097/ALN.0000000000003510. No abstract available. PMID 32833387
- [Background] Ramirez MF, Cata JP. Anesthetic care influences long-term outcomes: What is the evidence? Best Pract Res Clin Anaesthesiol. 2021 Dec;35(4):491-505. doi: 10.1016/j.bpa.2021.01.004. Epub 2021 Feb 3. PMID 34801212
- [Background] Allaire M, Goumard C, Lim C, Le Cleach A, Wagner M, Scatton O. New frontiers in liver resection for hepatocellular carcinoma. JHEP Rep. 2020 Jun 4;2(4):100134. doi: 10.1016/j.jhepr.2020.100134. eCollection 2020 Aug. PMID 32695968
- [Background] Asrani SK, Devarbhavi H, Eaton J, Kamath PS. Burden of liver diseases in the world. J Hepatol. 2019 Jan;70(1):151-171. doi: 10.1016/j.jhep.2018.09.014. Epub 2018 Sep 26. PMID 30266282